CLINICAL TRIAL: NCT03867214
Title: Effects of Oral Care With Glutamine on Oral Health, Oral Flora and Incidence of Pneumonia After Neurosurgery With Microbiome Analysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanzhao (Other)
Responsible Party: Sponsor-Investigator, Yanzhao, Dr, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJODCT2014003
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Oral Mucositis; Pneumonia
MeSH Terms: conditions — Stomatitis; Pneumonia | interventions — Glutamine; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): Receiving TXA, Study group
  Tranexamic acid, Study group tranexamic acid 1g,
  intravenous injection, pre-operationally
  Interventions: Drug: Glutamine
- Placebo Comparator (Placebo Comparator): Normal saline, Control group
  Not receiving tranexamic acid, Control group Normal
  saline 100mL, intravenous injection, pre-operationally
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Glutamine — 1 g of tranexamic acid in 100 mL of normal saline intravenously approximately 15 minutes before incision
  Arms: Experimental
Drug: Normal saline — 100 mL of normal saline intravenously approximately 15 minutes before incision
  Arms: Placebo Comparator

SUMMARY:
A randomized, double-blind, single-center and controlled study comparing the efficacy and safety of intravenous administration of tranexamic acid to reduce blood loss in simultaneous bilateral total knee arthroplasty.

DETAILED DESCRIPTION:
A randomized, double-blind, single-center and controlled study comparing the efficacy and safety of intravenous administration of tranexamic acid to reduce blood loss in simultaneous bilateral total knee arthroplasty. Subjects will be monitored for occurrence of any complications, particularly deep venous thrombosis and thromboembolism during the hospital stay and for 1 months postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who plan to undergo simultaneous primary total knee arthroplasty on bilateral knee joint with a diagnosis of osteoarthritis or aseptic bone necrosis, but not of rheumatoid arthritis;
* All patients who have normal preoperative platelet count, normal prothrombin time, normal partial thromboplastin time, and normal international normalized ratio;
* The use of only balanced electrolyte solutions and/or albumin for plasma volume restitution.

Exclusion Criteria:

* Allergy to tranexamic acid;
* Receiving warfarin or heparin; had a history of hemophilia, deep venous thrombosis, pulmonary embolism, or renal impairment; or were pregnant;
* Patients with any cardiovascular problems (such as myocardiac infarction history, atrial fibrillation, angina);
* Patients with thromboembolic disorders, or those exhibiting a deteriorating general condition;
* Preoperative anemia (a hemoglobin value of <11 g/dL in females and <12 g/dL in males), refusal of blood products;
* Preoperative use of anticoagulant therapy within five days before surgery, fibrinolytic disorders requiring intraoperative antifibrinolytic treatment, coagulopathy (as identified by a preoperative platelet count of <150,000/mm3, an international normalized ratio of >1.4, or a prolonged partial thromboplastin time [>1.4 times normal]).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Allogeneic Blood Transfusion as a Measure of Efficacy | one week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qingsheng Zhu, Study Director — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, China

IPD SHARING:
Plan to Share IPD: No